CLINICAL TRIAL: NCT05418283
Title: Effects of 12-week Exercise Program on Sleep Quality and Fear of Death in Geriatric Individuals
Acronym: EXDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXDES
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Sleep Disorder; Depressive Disorder; Death; Physical Inactivity
Keywords: sleep disorder; fear of death; exercise; Elderly
MeSH Terms: conditions — Sleep Wake Disorders; Depressive Disorder; Death; Sedentary Behavior; Necrophobia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): 12-week aerobic exercise program will be applied (3/week)
  Interventions: Behavioral: Exercise
- Control (No Intervention): No intervention will be applied.

INTERVENTIONS:
Behavioral: Exercise — 1 hour of aerobic exercise will be applied 3 days a week for 12 weeks.
  Arms: Exercise

SUMMARY:
The aim of this study is to determine the effect of regular aerobic exercise program on tanatophobia and sleep quality in elderly individuals, and to evaluate the relationship between sleep disorder and fear of death.

DETAILED DESCRIPTION:
The effect of regular exercise programs on fear of death in elderly individuals is unknown. The aim of this study is to determine the effect of regular aerobic exercise program on tanatophobia and sleep quality in elderly individuals, and to evaluate the relationship between sleep disorder and fear of death.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over who volunteered to participate in the study,
* Conscious and without communication problems,
* No orthopedic injury that prevents walking
* Those who are physically inactive according to the International Physical Activity Assessment Questionnaire
* Those who have sufficient motivation to participate in the exercise program (will be evaluated by a one-on-one interview by the researchers)
* Being eligible to participate in an exercise program after a cardiac examination by a cardiologist (resting ECG and questioning of cardiac symptoms, further examinations such as exercise ECG test if necessary)

Exclusion Criteria:

* Having a history of neuromuscular disease
* Serious medical condition (eg advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.) that would prevent the person from participating in exercise training.
* Less than 1 year life expectancy
* Having an orthopedic injury that prevents walking
* Presence of advanced sensory deficit
* Having visual and hearing problems
* Not having sufficient communication skills (Mini Mental Test score below 24 points)
* Not having agreed to participate in the study
* Uncontrolled hypertension
* Not being found suitable for exercise in the examination performed by physicians and physiotherapists

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
thanatophobia | 1 week
  evaluation of thanatophobia

SECONDARY OUTCOMES:
sleep quality | 1 week
  evaluation of sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Training And Research Hospital
Locations (1):
- Sultan Abdülhamid Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No